CLINICAL TRIAL: NCT03338023
Title: A Prospective, Randomized, Open-Label Comparison of a Long-Acting Basal Insulin Analog, LY2963016, to Lantus® in Combination With Mealtime Insulin Lispro in Adult Chinese Patients With Type 1 Diabetes Mellitus
Brief Title: A Study of LY2963016 Compared to Lantus® in Adult Chinese Participants With Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16036; I4L-GH-ABES (Other: Eli Lilly and Company)
Record Dates: First submitted 2017-11-07; First posted 2017-11-09 (Actual); Results first posted 2021-03-29 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2020-04-15

CONDITIONS: Type 1 Diabetes
Keywords: Insulin Glargine
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — LY2963016 insulin glargine; Insulin Glargine; Insulin Lispro

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- LY2963016 + Insulin Lispro (Experimental): Participants received 100 units per milliliter (U/mL) LY2963016 administered subcutaneously (SC) once daily (QD) and 100 U/mL premeal insulin lispro administered SC thrice-daily (TID) within 15 minutes before meals or immediately after the meal.
  Interventions: Drug: LY2963016; Drug: Insulin Lispro
- Lantus® + Insulin Lispro (Active Comparator): Participants received 100 U/mL Lantus® administered SC QD and 100 U/mL premeal insulin lispro administered SC thrice-daily (TID) within 15 minutes before meals or immediately after the meal.
  Interventions: Drug: Lantus®; Drug: Insulin Lispro

INTERVENTIONS:
Drug: LY2963016 — Administered SC
  Arms: LY2963016 + Insulin Lispro
Drug: Lantus® — Administered SC
  Arms: Lantus® + Insulin Lispro
Drug: Insulin Lispro — Administered SC

SUMMARY:
The purpose of this study is to compare long-acting basal insulin analog LY2963016 to Lantus® in combination with mealtime insulin lispro in adult Chinese participants with Type 1 Diabetes Mellitus (T1DM).

ELIGIBILITY:
Inclusion Criteria:

* Have T1DM based on the disease diagnostic criteria (World Health Organization [WHO] Classification).
* Have duration of T1DM ≥1 year.
* Have HbA1c ≤11 %.
* Have been administered with basal-bolus insulins or pre-mixed insulins for at least 90 days prior to screening.
* Have a body mass index (BMI) ≤35 kilograms per meter squared.

Exclusion Criteria:

* Exposure to an insulin glargine other than Lantus® within previous 30 days.
* Have had more than one episode of severe hypoglycemia within 6 months prior to entry into the study.
* Have had more than one episode of diabetic ketoacidosis or emergency room visits for uncontrolled diabetes leading to hospitalization within 6 months prior to entry into the study.
* Have known hypersensitivity or allergy to any of the study insulins (Lantus® or insulin lispro) or to excipients of the study insulins.
* Are pregnant, intend to become pregnant during the course of the study.
* Women who are breastfeeding.
* Are currently taking traditional medicine (herbal medicine or patent medicine) with known/specified content of anti-hyperglycemic effects within 3 months before screening.
* Have congestive heart failure Class III and IV.
* Have obvious clinical signs or symptoms, or laboratory evidence, of liver disease.
* Have any active cancer.
* Have a history or diagnosis of human immunodeficiency virus (HIV) infection.
* Have presence of clinically significant gastrointestinal disease.
* Have a history of renal transplantation, or are currently receiving renal dialysis.
* Are receiving chronic systemic glucocorticoid therapy at pharmacological doses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2018-03-23 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2020-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (20):
- China (20):
  - Peking University Peoples Hospital, Beijing, Beijing Municipality
  - Guangdong Province People's Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital, Sun-Yat Sen University, Guangzhou, Guangdong
  - Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Shantou University Medical College No.2 Affiliated Hospital, Shantou, Guangdong
  - The 1st Affiliated Hospital of Henan Science and technology, Luoyang, Henan
  - Wu Han Tongji Hospital, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Changzhou No.2 People's Hospital, Changzhou, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Nanjing First Hospital, Nanjing, Jiangsu
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - No.2 Hospital Affiliated to Jilin University, Changchun, Jilin
  - Dalian Med. Univ. No 2 Affiliate Hospital, Dalian, Liaoning
  - The First Affiliated Hospital with Nanjing Medical Universit, Nanjing, Nanjing
  - Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - First People's Hospital of Yunnan Province, Kunming, Yunnan
  - Peking Union Medical College Hospital, Beijing
  - Shanghai Putuo District Center Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and asigned data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Yan X, Feng C, Lou Y, Zhou Z. Efficacy and Safety of LY2963016 Insulin Glargine in Chinese Patients with Type 1 Diabetes Previously Treated with Insulin Glargine (Lantus(R)): a Post Hoc Analysis of a Randomized, Open-Label, Phase 3 Trial. Diabetes Ther. 2022 Jun;13(6):1161-1174. doi: 10.1007/s13300-022-01262-8. Epub 2022 Apr 26. PMID 35471721

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LY2963016 + Insulin Lispro | Lantus® + Insulin Lispro
Started | 137 | 135
Received at Least One Dose of Study Drug | 137 | 135
Completed | 128 | 125
Not Completed | 9 | 10
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Protocol Violation | 3 | 3
Not completed — Lost to Follow-up | 2 | 1
Not completed — Physician Decision | 1 | 2

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | LY2963016 + Insulin Lispro | Lantus® + Insulin Lispro | Total
Number analyzed (Participants) | 137 | 135 | 272
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.8 (15.0) | 41.4 (13.8) | 41.6 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 66 | 143
  Male | 60 | 69 | 129
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 137 | 135 | 272
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 137 | 135 | 272
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 137 | 135 | 272
Hemoglobin A1c (HbA1c) at Baseline [Mean (Standard Deviation); unit: Percentage of HbA1c] | 7.90 (1.32) | 7.85 (1.48) | 7.88 (1.40)
Duration of Diabetes in years [Mean (Standard Deviation); unit: years] | 10.29 (9.53) | 10.53 (9.53) | 10.41 (9.51)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per meter square (kg/m²)] | 21.90 (2.54) | 22.03 (2.32) | 21.96 (2.43)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c) (LY2963016 Noninferior to Lantus®)
Description: HbA1c is a form of hemoglobin that is measured primarily to identify the average plasma glucose concentration over prolonged periods of time. Least square (LS) mean was calculated using mixed-effects model for repeated measures (MMRM) with variables baseline HbA1c + Treatment + Pre-study treatment + Pre-study metformin or acarbose usage + Time + Time*Treatment (Type III sum of squares).
Time Frame: Baseline, Week 24
Population: All randomized participants who received at least one dose of study drug and had a baseline and postbaseline HbA1c value.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | LY2963016 + Insulin Lispro | Lantus® + Insulin Lispro
Number analyzed (Participants) | 127 | 125
Percentage of HbA1c | -0.20 (0.071) | -0.08 (0.071)
Statistical Analysis 1: Comparison: Lantus® + Insulin Lispro; Test type: Non-Inferiority — Noninferiority of LY2963016 to Lantus® was demonstrated at the 0.4% noninferiority margin and over 80 percent power; Mean Difference (Net) = -0.12, 95% CI 2-sided [-0.32 to 0.08]

2. Secondary Outcome: Change From Baseline in HbA1c (Lantus® Noninferior to LY2963016)
Description: HbA1c is a form of hemoglobin that is measured primarily to identify the average plasma glucose concentration over prolonged periods of time. LS mean was calculated using MMRM with variables baseline HbA1c + Treatment + Pre-study treatment + Pre-study metformin or acarbose usage + Time + Time*Treatment (Type III sum of squares).
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | LY2963016 + Insulin Lispro | Lantus® + Insulin Lispro
Number analyzed (Participants) | 127 | 125
Percentage of HbA1c | -0.20 (0.071) | -0.08 (0.071)
Statistical Analysis 1: Comparison: LY2963016 + Insulin Lispro vs Lantus® + Insulin Lispro; Test type: Non-Inferiority — Noninferiority of Lantus® to LY2963016 was demonstrated at the 0.4% noninferiority margin; Mean Difference (Net) = -0.12, 95% CI 2-sided [-0.32 to 0.08]

3. Secondary Outcome: Change From Baseline in 7-Point Self-Monitored Blood Glucose (SMBG) Values
Description: The self-monitored plasma glucose (SMBG) data were collected at the following 7 time points: Before Morning Meal Glucose, 2 Hours After Morning Meal Glucose, Before Mid-Day Meal Glucose, 2 Hours After Mid-Day Meal Glucose, Before Evening Meal Glucose, Bedtime Glucose and 0300 Am Glucose. LS mean was calculated using MMRM with variables Baseline + Pre-study Treatment + Pre-study Metformin or Acarbose Usage + HbA1c at Baseline + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, Week 24
Population: All randomized participants who received at least one dose of study drug and had a baseline and postbaseline SMBG value.
Measure: Least Squares Mean (Standard Error); unit: milligrams per deciliter (mg/dL)
Arm/Group | LY2963016 + Insulin Lispro | Lantus® + Insulin Lispro
Number analyzed (Participants) | 127 | 124
milligrams per deciliter (mg/dL)
  Before Morning Meal Glucose | -7.2 (3.64) | -0.4 (3.68)
  2 Hours After Morning Meal Glucose | -10.6 (4.77) | -2.8 (4.83)
  Before Mid-Day Meal Glucose | -4.6 (4.13) | 8.5 (4.21)
  2 Hours After Mid-Day Meal Glucose | -1.6 (4.76) | 1.9 (4.76)
  Before Evening Meal Glucose | -6.2 (4.78) | 4.8 (4.85)
  Bedtime Glucose | -0.4 (4.99) | 5.0 (5.06)
  0300 Am Glucose | -4.9 (3.87) | 2.5 (3.94)
Statistical Analysis 1: Comparison: LY2963016 + Insulin Lispro vs Lantus® + Insulin Lispro; Before Morning Meal Glucose; Test type: Superiority; p = 0.191, Mixed Models Analysis; Mean Difference (Net) = -6.8, 95% CI 2-sided [-17.0 to 3.4]
Statistical Analysis 2: Comparison: LY2963016 + Insulin Lispro vs Lantus® + Insulin Lispro; 2 Hours After Morning Meal Glucose; Test type: Superiority; p = 0.250, Mixed Models Analysis; Mean Difference (Net) = -7.8, 95% CI 2-sided [-21.2 to 5.5]
Statistical Analysis 3: Comparison: LY2963016 + Insulin Lispro vs Lantus® + Insulin Lispro; Before Mid-Day Meal Glucose; Test type: Superiority; p = 0.028, Mixed Models Analysis; Mean Difference (Net) = -13.1, 95% CI 2-sided [-24.7 to -1.5]
Statistical Analysis 4: Comparison: LY2963016 + Insulin Lispro vs Lantus® + Insulin Lispro; 2 Hours After Mid-Day Meal Glucose; Test type: Superiority; p = 0.599, Mixed Models Analysis; Mean Difference (Net) = -3.6, 95% CI 2-sided [-16.8 to 9.7]
Statistical Analysis 5: Comparison: LY2963016 + Insulin Lispro vs Lantus® + Insulin Lispro; Before Evening Meal Glucose; Test type: Superiority; p = 0.109, Mixed Models Analysis; Mean Difference (Net) = -11.0, 95% CI 2-sided [-24.4 to 2.5]
Statistical Analysis 6: Comparison: LY2963016 + Insulin Lispro vs Lantus® + Insulin Lispro; Bedtime Glucose; Test type: Superiority; p = 0.452, Mixed Models Analysis; Mean Difference (Net) = -5.4, 95% CI 2-sided [-19.4 to 8.6]
Statistical Analysis 7: Comparison: LY2963016 + Insulin Lispro vs Lantus® + Insulin Lispro; 0300 Am Glucose; Test type: Superiority; p = 0.180, Mixed Models Analysis; Mean Difference (Net) = -7.4, 95% CI 2-sided [-18.3 to 3.5]

4. Secondary Outcome: Percentage of Participants With HbA1c <7%
Description: HbA1c is a form of hemoglobin that is measured primarily to identify the average plasma glucose concentration over prolonged periods of time.
Time Frame: Week 24
Population: All randomized participants who received at least one dose of study drug and had baseline and postbaseline HbA1c value.
Measure: Number; unit: percentage of participants
Arm/Group | LY2963016 + Insulin Lispro | Lantus® + Insulin Lispro
Number analyzed (Participants) | 127 | 125
percentage of participants | 30.7 | 32.8
Statistical Analysis 1: Comparison: LY2963016 + Insulin Lispro vs Lantus® + Insulin Lispro; Test type: Superiority; p = 0.787, Fisher Exact

5. Secondary Outcome: Percentage of Participants With HbA1c ≤6.5%
Description: as for outcome 4
Time Frame: Week 24
Population: All randomized participants who received at least one dose of study drug and had baseline and postbaseline HbA1c value.
Measure: Number; unit: percentage of participants
Arm/Group | LY2963016 + Insulin Lispro | Lantus® + Insulin Lispro
Number analyzed (Participants) | 127 | 125
percentage of participants | 15.7 | 22.4
Statistical Analysis 1: Comparison: LY2963016 + Insulin Lispro vs Lantus® + Insulin Lispro; Test type: Superiority; p = 0.201, Fisher Exact

6. Secondary Outcome: Change From Baseline in Intrapatient Blood Glucose (BG) Variability, Measured by the Standard Deviation of 7-point SMBG
Description: Change From Baseline in Intrapatient blood glucose (BG). LS mean was calculated using MMRM with variables Baseline + Pre-study Treatment + Pre-study Metformin or Acarbose Usage + HbA1c at Baseline + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, Week 24
Population: All randomized participants who received at least one dose of study drug and had a baseline and postbaseline SMBG value.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | LY2963016 + Insulin Lispro | Lantus® + Insulin Lispro
Number analyzed (Participants) | 122 | 119
mg/dL | -2.9 (1.33) | -2.6 (1.34)
Statistical Analysis 1: Comparison: LY2963016 + Insulin Lispro vs Lantus® + Insulin Lispro; Test type: Superiority; p = 0.885, Mixed Models Analysis; Mean Difference (Net) = -0.3, 95% CI 2-sided [-0.4 to 3.4]

7. Secondary Outcome: Change From Baseline in Glycemic Variability of Fasting Blood Glucose
Description: Change From Baseline in Glycemic Variability of Fasting Blood Glucose. LS mean was calculated using MMRM with variables Baseline + Pre-study Treatment + Pre-study Metformin or Acarbose Usage + HbA1c at Baseline + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, Week 24
Population: All randomized participants who received at least one dose of study drug and had a baseline and postbaseline SMBG value.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | LY2963016 + Insulin Lispro | Lantus® + Insulin Lispro
Number analyzed (Participants) | 122 | 119
mg/dL
  Morning Pre-meal Standard Deviation | -9.0 (2.53) | -5.5 (2.56)
  Daily Mean Standard Deviation | -10.4 (1.69) | -8.6 (1.71)
Statistical Analysis 1: Comparison: LY2963016 + Insulin Lispro vs Lantus® + Insulin Lispro; Morning Pre-meal Standard Deviation; Test type: Superiority; p = 0.328, Mixed Models Analysis; Mean Difference (Net) = -3.5, 95% CI 2-sided [-10.6 to 3.6]
Statistical Analysis 2: Comparison: LY2963016 + Insulin Lispro vs Lantus® + Insulin Lispro; Daily Mean Standard Deviation; Test type: Superiority; p = 0.467, Mixed Models Analysis; Mean Difference (Net) = -1.7, 95% CI 2-sided [-6.5 to 3.0]

8. Secondary Outcome: Change From Baseline in Basal Insulin Dose
Description: Change from baseline in basal insulin dose. LS mean was calculated using MMRM with variables Baseline + Pre-study Treatment + Pre-study Metformin or Acarbose Usage + HbA1c at Baseline + Treatment + Time + Treatment*Time (Type III sum of squares). Variance-Covariance structure (Actual Measurement) = Unstructured. Variance-Covariance structure (Change from Baseline) = Unstructured.
Time Frame: Baseline, Week 24
Population: All randomized participants who received at least one dose of study drug and had a baseline and postbaseline Basal Insulin dose value.
Measure: Least Squares Mean (Standard Error); unit: Units per Day (U/day)
Arm/Group | LY2963016 + Insulin Lispro | Lantus® + Insulin Lispro
Number analyzed (Participants) | 129 | 127
Units per Day (U/day) | 0.7 (0.33) | 1.5 (0.33)
Statistical Analysis 1: Comparison: LY2963016 + Insulin Lispro vs Lantus® + Insulin Lispro; Test type: Superiority; p = 0.090, Mixed Models Analysis; Mean Difference (Net) = -0.8, 95% CI 2-sided [-1.7 to 0.1]

9. Secondary Outcome: Change From Baseline in Prandial Insulin Dose
Description: Prandial Insulin Dose. LS mean was calculated using MMRM with variables Baseline + Pre-study Treatment + Pre-study Metformin or Acarbose Usage + HbA1c at Baseline + Treatment + Time + Treatment*Time (Type III sum of squares). Variance-Covariance structure (Actual Measurement) = Unstructured. Variance-Covariance structure (Change from Baseline) = Unstructured.
Time Frame: Baseline, Week 24
Population: All randomized participants who received at least one dose of study drug and had a baseline and postbaseline Prandial Insulin dose value.
Measure: Least Squares Mean (Standard Error); unit: U/day
Arm/Group | LY2963016 + Insulin Lispro | Lantus® + Insulin Lispro
Number analyzed (Participants) | 129 | 127
U/day | 0.2 (0.49) | 1.4 (0.50)
Statistical Analysis 1: Comparison: LY2963016 + Insulin Lispro vs Lantus® + Insulin Lispro; Test type: Superiority; p = 0.089, Mixed Models Analysis; Mean Difference (Net) = -1.2, 95% CI 2-sided [-2.6 to 0.2]

10. Secondary Outcome: Change From Baseline in Body Weight
Description: Change from baseline in body weight. LS mean was calculated using MMRM with variables Baseline + Pre-study Treatment + Pre-study Metformin or Acarbose Usage + HbA1c at Baseline + Treatment + Time + Treatment*Time (Type III sum of squares). Variance-Covariance structure (Actual Measurement) = Unstructured. Variance-Covariance structure (Change from Baseline) = Unstructured.
Time Frame: Baseline, Week 24
Population: All randomized participants who received at least one dose of study drug and had a baseline and postbaseline weight value.
Measure: Least Squares Mean (Standard Error); unit: kilograms (kg)
Arm/Group | LY2963016 + Insulin Lispro | Lantus® + Insulin Lispro
Number analyzed (Participants) | 128 | 125
kilograms (kg) | 0.8 (0.21) | 0.9 (0.22)
Statistical Analysis 1: Comparison: LY2963016 + Insulin Lispro vs Lantus® + Insulin Lispro; Test type: Superiority; p = 0.770, Mixed Models Analysis; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.7 to 0.5]

11. Secondary Outcome: Change From Baseline in Insulin Treatment Satisfaction Questionnaire (ITSQ)
Description: The ITSQ is a validated 22-item questionnaire that was used to assess treatment satisfaction. Items were measured on a 7-point scale, with lower scores reflecting better outcomes. In addition to an overall score, scores were also obtained for 5 domains, including inconvenience of regimen, lifestyle flexibility, glycemic control, hypoglycemic control, and insulin delivery device. Raw domain and overall scores were transformed on a scale from 0 to 100, where a higher score indicated better treatment satisfaction.
  LS mean was calculated using ANCOVA with variables Baseline + Pre-study Treatment + Pre-study Metformin or Acarbose Usage + HbA1c at Baseline + Treatment (Type III sum of squares).
Time Frame: Baseline, Week 24
Population: All randomized participants who received at least one dose of study drug and had a baseline and postbaseline ITSQ score.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | LY2963016 + Insulin Lispro | Lantus® + Insulin Lispro
Number analyzed (Participants) | 130 | 131
score on a scale
  ITSQ Inconvenience of Regimen Transformed Score | 3.5 (1.30) | 3.8 (1.29)
  ITSQ Lifestyle Flexibility Transformed Score | 1.3 (1.86) | 2.0 (1.86)
  ITSQ Hypoglycemic Control Transformed Score | 3.2 (1.39) | 3.8 (1.38)
  ITSQ Glycemic Control Transformed Score | 6.9 (1.64) | 6.0 (1.64)
  ITSQ Insulin Delivery Device Satisfaction Transformed Score | 3.3 (1.26) | 2.9 (1.26)
  ITSQ Total Transformed Score | 3.3 (1.10) | 4.1 (1.10)
Statistical Analysis 1: Comparison: LY2963016 + Insulin Lispro vs Lantus® + Insulin Lispro; ITSQ Inconvenience of Regimen Transformed Score; Test type: Superiority; p = 0.879, ANCOVA; Mean Difference (Net) = -0.3, 95% CI 2-sided [-3.9 to 3.3]
Statistical Analysis 2: Comparison: LY2963016 + Insulin Lispro vs Lantus® + Insulin Lispro; ITSQ Lifestyle Flexibility Transformed Score; Test type: Superiority; p = 0.788, ANCOVA; Mean Difference (Net) = -0.7, 95% CI 2-sided [-5.9 to 4.5]
Statistical Analysis 3: Comparison: LY2963016 + Insulin Lispro vs Lantus® + Insulin Lispro; ITSQ Hypoglycemic Control Transformed Score; Test type: Superiority; p = 0.775, ANCOVA; Mean Difference (Net) = -0.6, 95% CI 2-sided [-4.5 to 3.3]
Statistical Analysis 4: Comparison: LY2963016 + Insulin Lispro vs Lantus® + Insulin Lispro; ITSQ Glycemic Control Transformed Score; Test type: Superiority; p = 0.681, ANCOVA; Mean Difference (Net) = 1.0, 95% CI 2-sided [-3.6 to 5.6]
Statistical Analysis 5: Comparison: LY2963016 + Insulin Lispro vs Lantus® + Insulin Lispro; ITSQ Insulin Delivery Device Satisfaction Transformed Score; Test type: Superiority; p = 0.819, ANCOVA; Mean Difference (Net) = 0.4, 95% CI 2-sided [-3.1 to 3.9]
Statistical Analysis 6: Comparison: LY2963016 + Insulin Lispro vs Lantus® + Insulin Lispro; ITSQ Total Transformed Score; Test type: Superiority; p = 0.605, ANCOVA; Mean Difference (Net) = -0.8, 95% CI 2-sided [-3.9 to 2.3]

12. Secondary Outcome: Number of Participants With Detectable Anti-Glargine Antibodies
Description: Number of participants with detectable anti-glargine antibodies
Time Frame: Baseline through Week 24
Population: All participants who received at least one dose of study drug.Only participants with detected or non-detected insulin antibody levels at baseline and post-baseline were included in analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | LY2963016 + Insulin Lispro | Lantus® + Insulin Lispro
Number analyzed (Participants) | 136 | 134
Participants
  Detectable Anti-Glargine Antibodies | 76 | 68
  Detectable Cross Reactive Insulin Antibodies | 67 | 58
  Treatment Emergent Antibody Response (TEAR) | 42 | 35

13. Secondary Outcome: Rate of Documented Symptomatic Hypoglycemia
Description: Hypoglycemic episodes are defined as events that are associated with reported signs and symptoms of hypoglycemia and/or documented blood glucose (BG) concentrations of ≤70 mg/dL (3.9 mmol/L). The overall yearly rates (events/participant/year) of those hypoglycemic events, calculated as, for each participant, the number of episodes times 365.25 and then divided by the participants treatment duration, will be summarized, and analyzed by a Negative-binomial regression model with treatment as fixed effects and log of (patient's treatment duration/365.25) as an offset variable.
Time Frame: Baseline through Week 24
Population: All randomized participants who received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: events/participant/year
Arm/Group | LY2963016 + Insulin Lispro | Lantus® + Insulin Lispro
Number analyzed (Participants) | 137 | 135
events/participant/year | 12.6 (2.42) | 14.0 (2.64)

ADVERSE EVENTS:
Time Frame: Baseline Up To 28 Weeks
Description: All participants who received at least one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants at risk adjusted accordingly.
Arm/Group | LY2963016 + Insulin Lispro | Lantus® + Insulin Lispro
All-Cause Mortality (participants affected / at risk) | 0/137 | 0/135
Serious Adverse Events (participants affected / at risk) | 9/137 | 8/135
Other Adverse Events (participants affected / at risk) | 84/137 | 77/135
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | LY2963016 + Insulin Lispro (N=137) | Lantus® + Insulin Lispro (N=135)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Diabetic retinopathy (Eye disorders) | 1 (1) | 0 (0)
Diabetic gastroenteropathy (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 3 (4)
Diabetic neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Hypoglycaemic coma (Nervous system disorders) | 1 (1) | 0 (0)
Nephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Perinephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1)
Ovarian disorder (Reproductive system and breast disorders) | 1/77 (1) | 0/66 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | LY2963016 + Insulin Lispro (N=137) | Lantus® + Insulin Lispro (N=135)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Palpitations (Cardiac disorders) | 0 (0) | 2 (2)
Diabetic retinopathy (Eye disorders) | 3 (3) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 2 (3) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 7 (9) | 3 (4)
Toothache (Gastrointestinal disorders) | 2 (2) | 6 (6)
Chest discomfort (General disorders) | 1 (1) | 2 (2)
Chest pain (General disorders) | 2 (2) | 1 (1)
Injection site haemorrhage (General disorders) | 2 (2) | 0 (0)
Injection site pain (General disorders) | 4 (4) | 7 (17)
Pyrexia (General disorders) | 1 (1) | 3 (3)
Hepatic function abnormal (Hepatobiliary disorders) | 2 (2) | 1 (1)
Hypersensitivity (Immune system disorders) | 2 (3) | 0 (0)
Bronchitis (Infections and infestations) | 4 (4) | 2 (2)
Conjunctivitis (Infections and infestations) | 2 (2) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 4 (4)
Influenza (Infections and infestations) | 3 (4) | 2 (2)
Nasopharyngitis (Infections and infestations) | 12 (15) | 14 (18)
Pharyngitis (Infections and infestations) | 1 (1) | 4 (5)
Upper respiratory tract infection (Infections and infestations) | 34 (43) | 23 (29)
Urinary tract infection (Infections and infestations) | 5 (5) | 2 (2)
Joint injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Thermal burn (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Blood creatinine increased (Investigations) | 2 (2) | 0 (0)
Blood urea increased (Investigations) | 2 (2) | 0 (0)
Platelet count decreased (Investigations) | 2 (2) | 1 (1)
Weight increased (Investigations) | 4 (4) | 4 (4)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3) | 3 (3)
Headache (Nervous system disorders) | 2 (2) | 2 (2)
Insomnia (Psychiatric disorders) | 3 (3) | 1 (1)
Azoospermia (Reproductive system and breast disorders) | 1/60 (1) | 0/69 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1/77 (1) | 0/66 (0)
Prostatitis (Reproductive system and breast disorders) | 1/60 (1) | 0/69 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Hypertension (Vascular disorders) | 4 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-03-02): https://cdn.clinicaltrials.gov/large-docs/23/NCT03338023/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-12): https://cdn.clinicaltrials.gov/large-docs/23/NCT03338023/SAP_001.pdf